



# Resource Optimization in the Intensive Care Unit Setting: A Staff Education and Scheduling Pilot Study to Improve Treatment Decisions and Staff Satisfaction

Minimal Risk Informed Consent Form for Participation in Educational Workshops

Study ID: 20200060-01 Version Date: 08/14/2020





#### Minimal Risk Informed Consent Form for Participation in Educational Workshops

**Study Title**: Resource Optimization in the Intensive Care Unit Setting: A Staff Education and Scheduling Pilot Study to Improve Treatment Decisions and Staff Satisfaction

**OHSN-REB Number**: 20200060-01H

Study Doctor: Kwadwo Kyeremanteng, Department of Critical Care, 613-789-5555, ext. 15072

Funder(s): Montfort Hospital Alternative Financing and Procurement and Ottawa's Department of

Medicine

# **INTRODUCTION**

You are being invited to participate in a pilot study for ICU staff designed to improve quality of care while reducing ICU costs, staff stress and burnout. Specifically, you are invited to participate and attend a series of educational workshops designed to increase clinicians' knowledge of cost-effective and evidence-based decision making about patient care (including tests, treatments and procedures) based on Choosing Wisely Canada recommendations. This consent form provides you with information to help you make an informed choice about the workshop. Please read this document carefully and ask any questions you may have. All your questions should be answered to your satisfaction before you decide whether to participate in this research study.

Please take your time in making your decision. You may find it helpful to discuss it with your friends, co-workers, and family.

Taking part in this study is voluntary. You have the option to not participate at all or you may choose to leave the study at any time. Whatever you choose, the decision will not affect your employment.

#### **IS THERE A CONFLICT OF INTEREST?**

There are no conflicts of interest to declare related to this study.

#### WHY IS THIS STUDY BEING DONE?

This is a pilot-study investigating ways to improve quality of care in the ICU through reducing ICU costs and reducing staff stress and burnout. The workshop you have chosen to participate in represents a step towards beginning a broader nationwide conversation on appropriate and evidence-centered care in Canadian ICU's. We hope this workshop will help empower you to make cost-effective and evidence-based decision-making about patient care when it comes to tests, treatments and procedures.

### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

It is difficult to anticipate the overall number of attendees in the workshops, but our aim is to make the workshops as accessible as possible to all interested ICU staff. Research sites include both the Civic and the General Campus' at The Ottawa Hospital and the Montfort Hospital in Ottawa.





This study should take about 12 months to complete, with a 3-month pre-intervention phase, a 6-month intervention phase, and a 3-month post-intervention phase. The results should be known in about 6 months from the end of the study.

## WHAT WILL HAPPEN DURING THIS STUDY?

#### Educational Workshop

You will be asked to attend one of several educational workshops offered throughout the 6-month intervention. The workshop will be facilitated by the study doctor (Dr. Kyeremanteng) a research assistant on the study team, and a medical student. The workshop will be approximately 2 to 3 hours in length depending on the level of participation and discussion among participants and will take place in a designated break room in the Intensive Care Units at each respective site. Throughout the workshop you will be given the opportunity to ask questions, express your opinion, give feedback and engage in general discussion about evidenced-based procedures, tests and treatments based on the Choosing Wisely Canada recommendations.

#### Post-workshop survey

A short survey will be handed out at the end of the workshop to evaluate the workshop and emailed the day after (in case you have to leave before the end of the workshop). The survey will take about 5-10 minutes to complete. A voluntary sign-up sheet will be circulated at the beginning of the workshop to collect some personal information including your name, title and email address. This information will solely be for the purpose of sending the post-educational workshop evaluation survey. The survey is completely voluntary, and your participation in the Educational workshop in no way requires that you participate in the evaluation.

The information you provide is for research purposes only. Some of the questions may be personal. You can choose not to answer questions if you wish.

# WHAT ARE THE RESPONSIBILITIES OF STUDY PARTICIPANTS?

If you choose to participate in this study, you will be expected to:

- Be present at the Educational workshop, however you may leave whenever you wish.
- Complete the voluntary evaluation survey
- Engage in discussion with your peers

#### **HOW LONG WILL PARTICIPANTS BE IN THE STUDY?**

Your participation on this study will only last for the duration of the workshop.

#### CAN PARTICIPANTS CHOOSE TO LEAVE THE STUDY?

You can choose to end your participation in this research (called withdrawal) at any time without having to provide a reason. If you choose to withdraw from the study, you are encouraged to contact the research team.

You may withdraw your permission to use information that was collected about you for this study at any time by letting the research team know. However, this would also mean that you withdraw from the study.





If you decide to leave the study, you can ask that the information that was collected about you not be used for the study. Let the research team know if you choose this.

#### WHAT ARE THE RISKS OR HARMS OF PARTICIPATING IN THIS STUDY?

There are no medical risks to you from participating in this study but taking part in this study may make you feel uncomfortable.

You may become uncomfortable while discussing your experiences. You may choose not to answer questions or leave the educational workshop at any time if you experience any discomfort.

#### WHAT ARE THE BENEFITS OF PARTICIPATING IN THIS STUDY?

We hope that from attending this workshop you will:

- Develop a better understanding of what common tests, procedures and treatments are unnecessary and could potentially be exposing patients to harm
- Gain some clear practical guidance for how to improve your practice and have conversations with your patients
- Contribute to improving educational initiatives for physicians

## HOW WILL PARTICIPANT INFORMATION BE KEPT CONFIDENTIAL?

If you decide to participate in this study, the research team will only collect the information they need for this study. A voluntary sign-up sheet will be circulated at the beginning of the workshop to collect your personal information including your name, title and email address. This information will be used solely for the purpose of sending out the post-educational workshop survey and will be destroyed immediately upon sending the follow up surveys.

We would like to note that communication via e-mail is not absolutely secure. We do not recommend that you communicate sensitive personal information via e-mail.

Records identifying you at this center will be kept confidential and, to the extent permitted by the applicable laws, will not be disclosed or made publicly available, except as described in this consent document.

Authorized representatives of the following organizations may look at your original (identifiable) records at the site where these records are held, to check that the information collected for the study is correct and follows proper laws and guidelines.

- The Ottawa Health Science Network Research Ethics Board who oversees the ethical conduct of this study.
- Ottawa Hospital Research Institute, to oversee the conduct of research at this location.

Information that is collected about you for the study (called study data) may also be sent to the organizations listed above. Your name, address, email, or other information that may directly identify you will not be used. The records received by these organizations may contain your study identification number.





If the results of this study are published, your identity will remain confidential. It is expected that the information collected during this study will be used in analyses and published to the scientific community at meetings and in journals.

Your de-identified data from this study may be used for other research purposes. If your study data is shared with other researchers, information that links your study data directly to you will not be shared.

Even though the likelihood that someone may identify you from the study data is very small, it can never be completely eliminated.

#### WHAT IS THE COST TO PARTICIPANTS?

Participation in this study will not involve any additional costs to you.

# ARE STUDY PARTICIPANTS PAID TO BE IN THIS STUDY?

You will not be paid for taking part in this study.

## WHAT ARE THE RIGHTS OF PARTICIPANTS IN A RESEARCH STUDY?

You will be told, in a timely manner, about new information that may be relevant to your willingness to stay in this study.

You have the right to be informed of the results of this study once the entire study is complete. If you would like to be informed of the results of this study, please let the study doctor know.

Your rights to privacy are legally protected by federal and provincial laws that require safeguards to ensure that your privacy is respected.

By signing this form, you do not give up any of your legal rights against the study doctor or involved institutions for compensation, nor does this form relieve the study doctor or their agents of their legal and professional responsibilities.

You will be given a copy of this signed and dated consent form prior to participating in this study.

#### WHOM DO PARTICIPANTS CONTACT FOR QUESTIONS?

If you have questions about taking part in this study you can talk to your study doctor, or the doctor who oversees the study at this institution. That person is:

Dr. Kwadwo Kyeremanteng
Principal Investigator Name

Telephone 613-263-0957

**Telephone** 

If you have questions about your rights as a participant or about ethical issues related to this study, you can talk to someone who is not involved in the study at all. Please contact The Ottawa Health Science Network Research Ethics Board, Chairperson at 613-798-5555 extension 16719.





**Study Title**: Resource Optimization in the Intensive Care Unit Setting: A Staff Education and Scheduling Pilot Study to Improve Treatment Decisions and Staff Satisfaction

## **SIGNATURES**

- All my questions have been answered,
- I understand the information within this informed consent form,
- I do not give up any of my legal rights by signing this consent form,
- I agree to take part in this study.

| Signature of Participant | Printed Name | Date | |
|--------------------------------|-----------------------|----------|---|
| Signature of Person Conducting | Printed Name and Role | <br>Date | _ |
| the Consent Discussion | Timed Name and Note | Date | |

Version date of this form: August 14, 2020